CLINICAL TRIAL: NCT05668728
Title: A Comparison for 3 Different Dry Needling Techniques for Myofacial Pain Syndrome Causing Servical Pain
Brief Title: Dry Needling for Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Emre Ata, Assoc Prof, Associate Proffesor, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2270
Record Dates: First submitted 2022-12-06; First posted 2022-12-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Myofascial Pain Syndromes; Neck Pain
Keywords: Dry Needling; Neck Pain; Myofascial Pain Syndromes
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain | interventions — spindlin

STUDY DESIGN:
Intervention Model Description: 3 GROUPS DİFFERENT TYPES OF DRY NEEDLİNG
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Dry needling + standard exercise program with 4 sessions of stick and pull out method at 1 week intervals
  Interventions: Other: Group 1: Peppering
- Group 2 (Active Comparator): Dry needling + standard exercise program with 4 sessions of turn-and-wait method at 1-week intervals
  Interventions: Other: group 2: spin and wait
- Group 3 (Active Comparator): Dry needling + standard exercise program with 4 sessions of stick and turn and wait method 1-week intervals
  Interventions: Other: group 3: Peppering and spin and wait

INTERVENTIONS:
Other: Group 1: Peppering — Before injection we will palpate the muscles of trapezius, m. rhomboideus, m. levator scapula for finding painful trigger points, and we will mark the point. the skin will be cleaned with an appropriate antiseptic. Before the needle is inserted, the area to be applied will be palpated once again to detect the painful trigger point between the thumb and index fingers. The needle will be guided to painful trigger points detected by palpation. Stainless steel 25x25 mm needles will be used for dry needling. The needle will be inserted and removed until the local twitch response disappears, at least 10 times at each point found. Afterwards, the patient will be given a standard exercise program for the neck muscles. With this method, dry needling will be applied to the patient 4 times a week, once a week.
  Arms: Group 1
Other: group 2: spin and wait — Just before the injection, painful trigger points in the bilateral muscles of trapezius, m. rhomboideus, and m. levator scapula will be identified and marked by palpation, and the skin will be cleaned with an appropriate antiseptic. Before the needle is inserted, the area to be applied will be palpated once again to detect the painful trigger point between the thumb and index fingers. The needle will be guided to painful trigger points detected by palpation. Stainless steel 25x25 mm needles will be used for dry needling. After the dry needle is inserted at each point found, it will be spinned counterclockwise and left. Waiting time for each patient will be limited to 15 minutes. Afterwards, the patient will be given a standard exercise program for the neck muscles. With this method, dry needling will be applied to the patient 4 times a week, once a week.
  Arms: Group 2
Other: group 3: Peppering and spin and wait — Just before the injection, painful trigger points in the bilateral muscles of trapezius, m. rhomboideus, and m. levator scapul will be identified and marked with palpation, and the skin will be cleaned with an appropriate antiseptic. Before the needle is inserted, the area to be applied will be palpated once again to detect the painful trigger point between the thumb and index fingers. The needle will be guided to painful trigger points detected by palpation. Stainless steel 25x25 mm needles will be used for dry needling. After the needle is inserted and removed, it will be spinned counterclockwise for 15 minutes in each patient until the local twitch response disappears, at least 10 times at each point found. Afterwards, the patient will be given a standard exercise program. With this method, dry needling will be applied to the patient 4 times a week, once a week.
  Arms: Group 3

SUMMARY:
Myofascial pain syndrome (MAS) is defined as a regional painful syndrome characterized by pain and tenderness in a muscle group or a muscle, a taut band within the muscle, pain reflected by pressing, and the presence of trigger points. It causes localized muscle pain in the shoulder and neck. The frequency of mas is around 12% in the normal population, and its frequency increases in those with chronic diseases. It is more common in the 30-60 age range and in the female population. Mechanical causes such as micro-macro trauma, nociceptive disorders, physical fatigue, psychological stress and genetic factors are blamed in its etiopathogenesis. Painful myofascial trigger points may occur by pressing on all muscles in the body, although it is more common in the trazius muscle, especially in those who work at a desk, who are constantly in a certain position, and who are sedentary. Myofascial trigger points are often detected by examination.

DETAILED DESCRIPTION:
There is a difference between the pain, neck extension range of motion, neck functional status of 3 different dry needling methods used in routine treatment in patients with myofascial pain syndrome. The investigators set out by thinking which method is more appropriate to choose in our practice. When the investigators examined the literature, the investigators could not find a study comparing these methods. However, at the points where sham needling, lidocaine administration, ozone cost, kinesiotaping methods and dry needling are compared by using these methods separately, regardless of the method of dry needling, there is a significant improvement in functional status, pain score, attachments, improvement expenses in the range of motion. However, the investigators think that it will contribute to a study literature on the protection of these purposes more clearly.

ELIGIBILITY:
Inclusion Criteria:

* Among the patients who applied to Sultan 2. Abdulhamid Han Hospital Physical Medicine and Rehabilitation Department and were diagnosed with myofascial pain syndrome
* Decided to receive dry needling treatment
* Between the ages of 18 and 65
* At least 1 painful myofascial trigger point in the m.trapezius, m.levator scapula muscles
* Patients with neck pain lasting less than 6 months

Exclusion Criteria:

* Those with a history of cervical operation
* Those who have a history of shoulder operation
* Patients with radiculopathy as a result of the examination
* Those who have been injected into the determined area in the last 3 months
* Those diagnosed with fibromyalgia according to the 2018 fibromyalgia scale
* Those with cervical disc herniation in the MR imaging taken within the last 1 year
* Pregnant/pregnant women
* Those who are allergic to silver
* Those with a history of malignancy
* Those with positive red flags
* Those with known rheumatological disease
* Those who do not accept dry needling
* Those with cognitive impairment
* Those who have local infection in the application area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Visuel Analog Scale | one month
  It is used to convert some values that cannot be measured numerically into numeric. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line, and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing. For example, for pain, I have no pain at one end and very severe pain at the other end, and the patient marks his/her current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain.

SECONDARY OUTCOMES:
Neck Disability Index | one month
  It is a questionnaire consisting of 10 questions and questions how neck pain affects the patient's ability to perform daily life activities such as sleep, personal care, driving, reading, and concentration. Each question is answered between 0-5 points. The minimum score can be 0, the maximum score can be 50. 0-4 points: no disability 5-14 points: mild disability 15-24 points: moderate disability 25-34 points: severe disability A score of 35 and above means complete disability
European Quality of Life 5 Dimensions 3 Level Version | One month
  It is a scale developed to evaluate health-related quality of life. It consists of two parts; one . The department defines the health profile in 5 dimensions (mobility, self-care, social life, pain, psychological state). Each dimension contains three statements according to the degree of difficulty (1: some problem, 2: moderate, 3: a lot of problems), the second part includes a visual analog scale (VAS) on which respondents rate their current health status from 0 to 100. It is easy to apply and is completed in a short time. 100 describes best functional stiuation, 0 describes worst developed to evaluate health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Ass.Prof., Principal Investigator — Sultan II. Abdulhamidhan Training and Research Hospital
Locations (1):
- Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stieven FF, Ferreira GE, Wiebusch M, de Araujo FX, da Rosa LHT, Silva MF. Dry Needling Combined With Guideline-Based Physical Therapy Provides No Added Benefit in the Management of Chronic Neck Pain: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2020 Aug;50(8):447-454. doi: 10.2519/jospt.2020.9389. Epub 2020 Apr 9. PMID 32272030
- [Result] Gattie E, Cleland JA, Snodgrass S. The Effectiveness of Trigger Point Dry Needling for Musculoskeletal Conditions by Physical Therapists: A Systematic Review and Meta-analysis. J Orthop Sports Phys Ther. 2017 Mar;47(3):133-149. doi: 10.2519/jospt.2017.7096. Epub 2017 Feb 3. PMID 28158962
- [Result] Raeissadat SA, Rayegani SM, Sadeghi F, Rahimi-Dehgolan S. Comparison of ozone and lidocaine injection efficacy vs dry needling in myofascial pain syndrome patients. J Pain Res. 2018 Jun 29;11:1273-1279. doi: 10.2147/JPR.S164629. eCollection 2018. PMID 29988746